CLINICAL TRIAL: NCT02076295
Title: [18F]Flubatine: a Novel Biomarker of Cholinergic a4ß2 Nicotinic Receptors and Cognition in Parkinson's Disease
Brief Title: Cholinergic Nicotinic Receptors and Cognition in PD
Acronym: CHONI
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Martijn Muller, Research Assistant Professor, University of Michigan
Other Study IDs: HUM00083054
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease
Keywords: Cognition; Cholinergic nicotinic receptors; Positron Emission Tomography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples to collect DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease subjects
- Normal control subjects

SUMMARY:
Mild cognitive impairment and dementia are frequent non-motor complications of moderate to advanced Parkinson's disease. Brain positron emission tomography (PET) study findings confirm post-mortem evidence that cholinergic loss is related to cognitive impairment in Parkinson's disease. However, current cholinergic augmentation therapy is not always effective and it should only target those Parkinson's disease patients who have evidence of cholinergic system impairment. The objective of this study is to study the association of a particular subtype of cholinergic receptors, so-called nicotinic acetylcholine receptors, with cognition in Parkinson's disease using a novel PET marker of cholinergic system integrity.

DETAILED DESCRIPTION:
Parkinson's disease patients will undergo nicotinic acetylcholine receptor PET imaging with the radioligand [18F]flubatine and MRI on one day and extensive neuropsychological testing on another day. The degree of nicotinic receptor expression obtained with PET imaging will be correlated with the neuropsychology test results.

Positive [18F]flubatine PET findings in this study would establish nicotinic receptors as an important contributor to cognitive dysfunction in Parkinson's disease and could kindle pharmaceutical interest in pursuing these agents for Parkinson's disease applications.

We expect that lower nicotinic receptor expression is associated with impaired cognitive functioning in Parkinson's disease. In a personalized medicine approach the PET radioligand [18F]flubatine could serve as an important marker to identify those patients who are expected to benefit most from nicotinic receptor drug treatment.

ELIGIBILITY:
Inclusion criteria:

* PD subjects (M/F, non-smoking, ≥ 50 years old, Hoehn & Yahr stages 1-4)
* Normal control subjects (N=15, M/F, non-smoking, ≥ 50 years old)

Exclusion Criteria:

* Active smoking, use of other tobacco products, or use of nicotinic drugs such as nicotine patches or varenicline.
* Subjects with contra-indications to MR imaging, including pacemakers or claustrophobia.
* Evidence of large vessel stroke or mass lesion on MRI.
* Use of (anti-)cholinergic or neuroleptic drugs.
* Dementia or severe cognitive impairment confirmed by clinical and detailed neuropsychological assessment precluding safe study participation, performing study procedures, or unable to follow directions by study personnel.
* Evidence of atypical parkinsonism on neurological exam.
* Subjects limited by participation in research procedures involving ionizing radiation.
* Pregnancy (test within 48 hours of each PET session) or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Primary care clinic
  * Community sample
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Cerebral cholinergic nicotinic receptor expression | Will be assessed during the neuroimaging study visit(s); typically 1 day
  Cortical and sub-cortical [18F]flubatine binding

SECONDARY OUTCOMES:
Cognitive performance | Will be assessed during the clinical visit(s); typically 1 day
  Composite score of cognitive performance

CONTACTS AND LOCATIONS:
Overall Officials: Martijn T Muller, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No